CLINICAL TRIAL: NCT01648881
Title: Dissection of Aorta: Descending Part, Imaging
Brief Title: Imaging of Dissection of the Descending Aorta
Acronym: DADI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P 100505; 2011-A00238-33 (Other: ID RCB)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Dissection of the Descending Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: TEP-18FDG for every patient after aortic dissection — Cover key details of the intervention. Must be sufficiently detailed to distinguish between arms of a study (e.g., comparison of different dosages of drug) and/or among similar interventions (e.g., comparison of multiple implantable cardiac defibrillators). For example, interventions involving drugs may include dosage form, dosage, frequency and duration.
  Example: 50 mg/m2, IV (in the vein) on day 5 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: TEP-18FDG

SUMMARY:
Patients with dissection of the descending aorta will be followed up according to a precise timeline.

DETAILED DESCRIPTION:
NMR baseline A PET Scanner will be performed minimum 3 months post dissection 6 months and every year during three years after PET scanner : CT scanner and blood sample

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Seen for dissection of the descending aorta
* Dissection of the descending aorta within the last three months
* Affiliation to social security
* Signed informed consent

Exclusion Criteria:

* intervention programmed in relation with dissection of the descending aorta
* Pregnant female
* Adults without legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dissection of the descending aorta
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume JONDEAU, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pr Guillaume JONDEAU . Cardiologie. Hôpital Bichat, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided